CLINICAL TRIAL: NCT04391088
Title: Evaluation of Vaccination Coverage in People Linving With Diabetes
Brief Title: Vaccination Coverage in People Linving With Diabetes
Acronym: VacDiab
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0575
Record Dates: First submitted 2020-05-12; First posted 2020-05-18 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-06

CONDITIONS: Diabetes
Keywords: People over 18 years old; vaccines; Diabetes; Clinical pharmacy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hospitalized people living with diabetes: hospitalized people living with diabetes
  Interventions: Other: vaccine coverage assessment

INTERVENTIONS:
Other: vaccine coverage assessment — vaccine coverage assessment

SUMMARY:
For several years, the prevalence of people living with diabetes (pDT) has been steadily increasing. It was estimated by the health insurance in 2016 at 5 %, or more than 3.3 million people in France. By different physiological mechanisms, diabetes is associated with immunodeficiency. As a result, several vaccines are recommended in pDT.

The vaccination policy is drawn up in France by the French Minister of Health, who makes public the vaccination schedule after the opinion of the High Authority of Health.

Currently according to the 2019 immunization schedule, the dTP vaccine is the only mandatory in the general population with recalls in adults aged 25, 45, 65 and every 10 years. This vaccine is especially indicated for this segment of the population because diabetes is a risk factor for tetanus. In 2011, the Ministry of Health estimated that only 50.5% of the general population was up to date against dTP.

Two vaccines are recommended for pDT according to the current vaccine schedule: the flu vaccine and the pneumococcal vaccine. In fact, influenza and pneumococcal disease are more frequent and more serious for these patients compared to the general population. Influenza vaccine has to be done annually in the early winter period. The vaccine coverage for winter 2018/2019 was estimated at 46.8 % of the target population. The vaccination scheme for pneumococcal vaccine is more complex: it involves a primary vaccination with a vaccine with 13 valences followed by another with 23 valences at least eight weeks later. Thereafter, a recall is to be carried out every five years with the 23 valences vaccine. Vaccination coverage was estimated in France in 2011 at 8.1 % in the population at risk.

According to several studies, the shingles virus has a greater impact and is more aggressive in pDT than in the general population. Similarly, the virus would tend to unbalance diabetes. There is currently a vaccine against shingles that is recommended and reimbursed in the population aged 65 to 74 years.

In our practice, a pharmaceutical team has been carrying out medication reconciliation for several years at the hospital admission and discharge of the patient in the endocrinology-nutrition department of the university hospital of Montpellier.

During this medication reconciliation, a pharmaceutical interview on the management of drug treatments is carried out . Since May 2019, we added to this interview an assessment of the vaccination coverage and feelings of people regarding vaccination. Following this assessment, a report is made during an interview with the doctor responsible for the patient. During this interview, the update of mandatory and recommended vaccinations are discussed between the doctor and the pharmacist.

In this context, it seems interesting to us to make an assessment of our practices and the investigator make the following assumptions:

* There is a defect in the mandatory and recommended process of vaccination for pDT
* A synthesis of pDT vaccine status between the physician and the pharmacist at the time of hospitalization would allow optimization of vaccine management in accordance with current recommendations and practices.

The main objective of the study is to assess vaccine coverage for mandatory and recommended pDT vaccines at hospital admission.

The secondary objectives are:

* Description of pDT experience with vaccination;
* Description of the management of vaccination within the Department of Endocrinology-Nutrition-Diabetes during and after the patient's hospitalization in terms of (intra-hospital vaccination, hospital prescriptions of a vaccine after hospitalization and number of vaccination recommendations in the hospitalization report).
* Description of transmission of vaccination status of patients to their treating physician

ELIGIBILITY:
Inclusion criteria:

* Patients aged above 18 years old,
* People living with diabetes

Exclusion criteria:

• Patients hospitalized for diabetes discovery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population was composed of people living with diabetes hospitalized in Diabetes-Nutrition unit of Montpellier University hospital
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
number of diabetic patients up to date with their mandatory and recommended vaccinations | 1 day (at hospital admission)
  number of diabetic patients up to date with their mandatory and recommended vaccinations

SECONDARY OUTCOMES:
number of patients vaccinated during hospitalization | 1 day (from the day of admission to the day of discharge)
  number of patients vaccinated during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Cyril BREUKER, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC